CLINICAL TRIAL: NCT05389345
Title: Effects of Adding Transcranial Direct Current Stimulation to Executive Function Training for Schizophrenia-spectrum Disorders - a Randomized Control Trial
Brief Title: tDCS and Executive Function Training for Schizophrenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not started.
Sponsor: University of Toronto (Other)
Collaborators: Ontario Shores Centre for Mental Health Sciences (Other)
Responsible Party: Principal Investigator, Michael Best, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41543
Record Dates: First submitted 2022-05-17; First posted 2022-05-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Schizophrenia Spectrum Disorder; Schizophrenia and Related Disorders
Keywords: Schizophrenia; Cognitive remediation; Transcranial direct current stimulation; tDCs; CR; cognitive rehabilitation; executive function training; ET
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation; Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either actual transcranial direct current stimulation (tDCS) or sham tDCS prior to engaging in executive function training (ET). All participants will receive ET.
Who Masked: Outcomes Assessor
Masking Description: The randomization sequence will be pre-generated by the study coordinator who will then inform the treating clinician. The assessors obtaining outcome measure data will be blind to participants' assigned treatment groups. Participants will not be told which stimulation group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual tDCs + ET (Experimental): All interventions will involve 4 weeks of group intervention consisting of two 1-hour group sessions per week and additional practice between sessions. Half of study participants will be randomized to receive 30 minutes of transcranial direct current stimulation (tDCS) prior to beginning each ET session. ET session will begin immediately after tDCS.
  Interventions: Behavioral: Transcranial direct current stimulation; Behavioral: Executive function training
- Sham tDCs + ET (Sham Comparator): All interventions will involve 4 weeks of group intervention consisting of two 1-hour group sessions per week and additional practice between sessions. Half of study participants will be randomized to receive 30 minutes of sham transcranial direct current stimulation (tDCS) prior to beginning each ET session. ET session will begin immediately after tDCS. During the sham tDCS, the procedures will be exactly the same as the real tDCS (e.g., application of electrodes), however, no stimulation will be provided when the device turned on.
  Interventions: Behavioral: Executive function training

INTERVENTIONS:
Behavioral: Transcranial direct current stimulation — Participants will receive bilateral prefrontal anodal stimulation with cathode placed on the back of the upper neck. Transcranial direct current stimulation (tDCS) will be delivered by a research assistant under the supervision of a psychiatrist.
  Other Names: tDCS
  Arms: Actual tDCs + ET
Behavioral: Executive function training — The Executive Training (ET) aspect of the study will be completed by all participants. ET sessions consist of 50% of the session practicing computerized cognitive training exercises, and 50% of the session developing cognitive strategies to use in the computerized exercises. Participants are encouraged to complete 40 minutes of computerized training per day, and complete strategy worksheets, on the unit or in the library at Ontario Shores between sessions. ET will be delivered virtually and group sessions will be conducted using the online platform Zoom. For any group sessions, a PHIPA and PIPEDA compliant license will be used. This means that participants will not be able to record their screen using Zoom or a third-party program. Dr. Best will also go through some rules during the first group Zoom session regarding the use of third-party equipment and the importance of confidentiality.
  Other Names: ET; Cognitive remediation; CR

SUMMARY:
Schizophrenia-spectrum disorders are the most persistent, debilitating, and economically burdensome mental illnesses worldwide. Cognitive remediation (CR) is a psychological intervention based on principles of learning and neuroplasticity to improve cognitive abilities. The investigators previously developed a novel CR intervention specifically targeting executive functions and aimed here to enhance its effect on functioning by combining it with Transcranial direct current stimulation (tDCs). The primary goal is to determine whether receiving tDCS prior to CR improves one's ability to engage in cognitive activities and enhance cognitive abilities. To do so, 40 participants will be recruited with schizophrenia-spectrum disorders from Ontario Shores inpatient units, half of whom will receive real tDCS and half will receive sham tDCS, whereas all will receive CR. This study will provide important information on whether the outcome of training executive function can be further enhanced with non-invasive brain stimulation.

DETAILED DESCRIPTION:
Schizophrenia-spectrum disorders are the most persistent, debilitating, and economically burdensome mental illnesses worldwide, and are associated with the greatest per-patient expense of all mental health conditions. Schizophrenia is associated with a 15-20 year decrease in life expectancy, 5-fold increase in likelihood of death by suicide, and a significant decrease in quality of life. Antipsychotic medications are the first line treatment for individuals with schizophrenia-spectrum disorders and are prescribed to nearly every service-user. However, in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) trial (one of the largest antipsychotic trials in 1493 individuals with schizophrenia), medication effects on psychosocial functioning were small (d = 0.25). Thus, the primary treatment available to all individuals with schizophrenia does little to improve community functioning. This may partially be a result of the limited efficacy of antipsychotic medication to improve neurocognitive abilities, widely recognized as a core feature of schizophrenia, and one recommendation stemming from the CATIE trial was that "more intensive psychosocial rehabilitative services, including cognitive rehabilitation, may be needed to affect more substantial gains in functioning."

Cognitive remediation (CR) is a psychological intervention based on principles of learning and neuroplasticity to improve neurocognitive abilities with the ultimate goal of improving community functioning. The neuroplastic effects of CR are well established with evidence for increased gray matter volume in the hippocampus and amygdala, increased activation of the medial prefrontal cortex, and increased amplitude of the mismatch negativity event-related potential following CR. In two recent randomized controlled trials (RCTs), we also demonstrated that CR improves synchronization of neural networks in the alpha and theta frequency bands. Meta-analyses support moderate transfer of these neurophysiological improvements to neurocognitive abilities (d = 0.45) and community functioning (d = 0.37). In a recent systematic review, we reported that CR approaches vary widely, but approaches that incorporate training of executive functions are generally the most effective. Based on these findings we developed a novel CR intervention specifically targeting executive functions and conducted two double-blind RCTs, in which targeted executive function training (ET) produced greater improvements in neurophysiology, neurocognition, functional skills and real-world community functioning compared to other leading forms of CR. This intervention is approximately half the duration of other CR programs, yet produces larger effect size improvements in community functioning.

Further augmentation of CR is needed to increase effect size and impact on community functioning in schizophrenia. One such augmentation strategy is via interventions that are known to enhance neuroplasticity, which is the underlying mechanism of learning. A promising neuroplasticity enhancing methodology is via non-invasive brain stimulation.

Transcranial direct current stimulation (tDCs) is the most common form of non-invasive transcranial electric stimulation (tES). Unlike other forms of transcranial electric stimulation (for example electroconvulsive therapy of ECT), tDCS is designed to modify cortical excitability by making underlying neurons more or less likely to fire but is not designed to induce depolarization or action potential in the neurons. tDCS involves application of a weak, constant (i.e., "direct") electric current from one electrode (anode) placed on the scalp to another (cathode) in order to modify cortical excitability. The application strength can be measured by amplitude of the current applied (usually one or two Amperes) and duration of application (usually around 20-30 minutes). tDCS is thought to be relatively safe with main side effect of local skin irritation and local skin burn. The risk of inducing a seizure is extremely low (mainly pediatric case report evidence), and in fact tDCS has literature support suggesting potentially anti-seizure effects. tDCS has been investigated for several therapeutic applications including cognitive disorders with promising results. There are some preliminary studies that support the feasibility, safety and promising efficacy of tDCS in combination with CR in schizophrenia. These studies are generally small and focused on cognitive domains such as working memory. More studies are needed to evaluate the added value of tDCS on effect size and impact on executive and community functioning.

Although cognitive remediation approaches such as ET improve community functioning for people with schizophrenia-spectrum disorders, these approaches may be further refined to improve efficacy. One option is to combine ET with neurostimulation designed to prime the brain for enhanced learning. In order to further increase the efficiency and effectiveness of ET it is necessary to determine whether receiving tDCS prior to engaging in this cognitive training intervention may enhance one's ability to engage in cognitive activities, or may improve their cognitive abilities. This will provide important information regarding whether the outcomes of ET can be further enhanced, which will directly inform clinical methods and optimize the effectiveness of this treatment.

The primary goal of this study is to:

(1) Examine the efficacy of combined Executive Training and tDCS compared to Executive Training combined with sham tDCS on neurocognition and functioning.

The participants for this study will be recruited from Ontario Shores inpatient units, specifically Complex General Psychiatry (CGP) inpatient units, which historically averages a length of stay of 51 to 159 days depending on the specific unit and typically comprises 70 to 75 patients at any given time with diagnoses of schizophrenia/schizophrenia spectrum disorders. Inpatients who are not expected to be discharged for 4 weeks (period needed for study interventions) will be enrolled. However, if a participant is discharged before the end of the treatment, arrangements will be made for him/her to complete the intervention by coming on-site daily for tDCS and ET.

Participants will be randomized using an online random number table to receive actual tDCS prior to engaging in ET or sham tDCS prior to engaging in ET. All participants will receive ET. The randomization sequence will be pre-generated by the study coordinator who will then inform the treating clinician. Three assessments will be completed over the course of the study: one within 1 to 2 weeks of the start of the intervention, one within 1 to 2 weeks after the intervention is complete, and one 3-months after the intervention is complete. Each assessment will last about 2.5 hours and can be conducted over two days according to participant preference. These assessments will involve paper/pencil tests and questionnaires, computerized tests, and Electroencephalogram (EEG) recordings.

Primary and secondary outcomes will be examined using Linear Mixed Models on the Intent-to-Treat sample with missing data interpolated using maximum likelihood estimation. The primary endpoint is the 3-month follow-up assessment, and secondary endpoint of post-intervention will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* those who meet the criteria of schizophrenia, schizoaffective disorder or any other psychotic disorder based on the DSM-V criteria
* 18-65 years of age
* know how to use a computer
* are not abusing drugs or alcohol (criteria met for abuse in the last month)
* can read and speak English

Exclusion Criteria:

* anyone enrolled in a cognitive training program in the last 6 months
* anyone with a neurological disease or neurological damage, medical illnesses that can change neurocognitive function, medical history of head injury with loss of consciousness
* with a neurological disease or neurological damage, medical illnesses that can change neurocognitive function, medical history of head injury with loss of consciousness
* those with a seizure disorder
* those who are pregnant
* those with psychotic symptoms that in the opinion of the study psychiatrist, would impose risk of distress and/or decompensation of psychosis (e.g. delusion of influence through electricity)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific Levels of Functioning (SLOF) | Change from baseline to 3-month follow-up
  The SLOF scale is a measure of community functioning

SECONDARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The CANTAB is a battery consisting of highly sensitive, precise and objective measures of cognitive function. It includes tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control.
Reading subtest of the Wide Range Achievement Test (WRAT) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The WRAT is an academic skills assessment which measures reading skills and provides an estimate of premorbid intellectual ability.
Questionnaire About the Process of Recovery (QPR) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The QPR was developed from service users' accounts of recovery from psychosis in collaboration with local service users. It asks people living with psychosis about aspects of recovery that are meaningful to them, and is strongly associated with general psychological wellbeing, quality of life and empowerment. This version contains 22 items while the response to each statement is scored on a 5-point Likert scale ranging from "0 = strongly disagree" to "4 = strongly agree". The lowest possible score is 0 and the highest score could be 88. Higher scores would indicate better recovery.
Brief Psychiatric Rating Scale (BPRS) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The BPRS measures psychopathology and symptom severity and is sensitive to changes in symptom levels
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The Q-LES-Q is a sensitive measure of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning.
Dysfunctional Attitudes Scale (DAS) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  DAS is a 40-item self-report measure assessing self-defeating attitudes theorized to underlie clinical depression and anxiety. The degree of agreement to each statement is scored on a 7-point Likert scale (1 = agree totally, 2 = agree very much, 3 = agree slightly, 4 = neutral, 5 = disagree slightly, 6 = disagree very much, 7 = disagree totally). The lowest possible scale is 40 while the highest possible scale is 280. Higher scores would indicate more negative beliefs.
Brief Core Schema Scale (BCSS) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The BCSS is a 24-item self-report measure assessing positive and negative judgments individuals hold about themselves and others. Responses are first given dichotomously as "no" or "yes". "No" is scored as 0 and if the answers are "yes", the intensity of beliefs are then rated on a 4-point scale (1 = believe it slightly, 2 = believe it moderately, 3 = believe it very much, 4 = believe it totally). The lowest score would be a 0 and the highest score would be a 96. Higher scores in the positive-self subscale indicate more positive beliefs about selves, while higher scores in the negative-self subscale indicate more negative beliefs about selves. Higher scores in the positive-others subscale indicate more positive beliefs about others, while higher scores in the negative-others subscale indicate more negative beliefs about others.
Generalized Self-Efficacy Scale (GSES) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The GSES assess optimistic self-beliefs to cope with a variety of difficult demands in life
Cognitive Failures Questionnaire (CFQ) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The CFQ was designed to measure perception, memory, and motor lapses in daily life
Need for Cognition Scale (NCS) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The NCS measures the tendency for an individual to engage in and enjoy thinking
Davos Assessment of Cognitive Biases (DACOBS) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The DACOBS is a 42-item self-report inventory measuring cognitive biases and discriminates between schizophrenia-spectrum patients and normal control subjects. The degree of agreement to each statement is scored on a 7-point Likert scale, ranging from "1 = strongly disagree" to "7 = strongly agree". The lowest score would be a 42 and the highest score would be a 294. Higher scores would indicate more cognitive biases.
Motivation and Pleasure Scale - Self-Report (MAP-SR) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  The MAP-SR assess the motivation and pleasure domains of negative symptoms.
Electroencephalogram (EEG) | baseline within 1-2 weeks of start of intervention, 1-2 week follow-up after intervention complete, 3-month follow up
  EEG will also be assessed using the Emotiv portable EEG system to assess neural synchronization to better understand how neural signatures change before and after the intervention. All EEG will be performed at Ontario Shores. Synchronization in the alpha and theta frequency bands during standard working memory and attention tests will be used to assess synchronization.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Best, PhD, Principal Investigator — University of Toronto
Locations (1):
- Ontario Shores Centre for Mental Health Sciences (Ontario Shores), Whitby, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu EQ, Birnbaum HG, Shi L, Ball DE, Kessler RC, Moulis M, Aggarwal J. The economic burden of schizophrenia in the United States in 2002. J Clin Psychiatry. 2005 Sep;66(9):1122-9. doi: 10.4088/jcp.v66n0906. PMID 16187769
- [Background] Palmer BA, Pankratz VS, Bostwick JM. The lifetime risk of suicide in schizophrenia: a reexamination. Arch Gen Psychiatry. 2005 Mar;62(3):247-53. doi: 10.1001/archpsyc.62.3.247. PMID 15753237
- [Background] Eack SM, Newhill CE. Psychiatric symptoms and quality of life in schizophrenia: a meta-analysis. Schizophr Bull. 2007 Sep;33(5):1225-37. doi: 10.1093/schbul/sbl071. Epub 2007 Jan 4. PMID 17204532
- [Background] Swartz MS, Perkins DO, Stroup TS, Davis SM, Capuano G, Rosenheck RA, Reimherr F, McGee MF, Keefe RS, McEvoy JP, Hsiao JK, Lieberman JA; CATIE Investigators. Effects of antipsychotic medications on psychosocial functioning in patients with chronic schizophrenia: findings from the NIMH CATIE study. Am J Psychiatry. 2007 Mar;164(3):428-36. doi: 10.1176/ajp.2007.164.3.428. PMID 17329467
- [Background] Eack SM, Hogarty GE, Cho RY, Prasad KM, Greenwald DP, Hogarty SS, Keshavan MS. Neuroprotective effects of cognitive enhancement therapy against gray matter loss in early schizophrenia: results from a 2-year randomized controlled trial. Arch Gen Psychiatry. 2010 Jul;67(7):674-82. doi: 10.1001/archgenpsychiatry.2010.63. Epub 2010 May 3. PMID 20439824
- [Background] Subramaniam K, Luks TL, Fisher M, Simpson GV, Nagarajan S, Vinogradov S. Computerized cognitive training restores neural activity within the reality monitoring network in schizophrenia. Neuron. 2012 Feb 23;73(4):842-53. doi: 10.1016/j.neuron.2011.12.024. PMID 22365555
- [Background] Best MW, Milanovic M, Iftene F, Bowie CR. A Randomized Controlled Trial of Executive Functioning Training Compared With Perceptual Training for Schizophrenia Spectrum Disorders: Effects on Neurophysiology, Neurocognition, and Functioning. Am J Psychiatry. 2019 Apr 1;176(4):297-306. doi: 10.1176/appi.ajp.2018.18070849. Epub 2019 Mar 8. PMID 30845819
- [Background] Best MW, Gale D, Tran T, Haque MK, Bowie CR. Brief executive function training for individuals with severe mental illness: Effects on EEG synchronization and executive functioning. Schizophr Res. 2019 Jan;203:32-40. doi: 10.1016/j.schres.2017.08.052. Epub 2017 Sep 19. PMID 28931460
- [Background] Wykes T, Spaulding WD. Thinking about the future cognitive remediation therapy--what works and could we do better? Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S80-90. doi: 10.1093/schbul/sbr064. PMID 21860051
- [Background] Best MW, Bowie CR. A review of cognitive remediation approaches for schizophrenia: from top-down to bottom-up, brain training to psychotherapy. Expert Rev Neurother. 2017 Jul;17(7):713-723. doi: 10.1080/14737175.2017.1331128. Epub 2017 May 24. PMID 28511562
- [Background] Zhao H, Qiao L, Fan D, Zhang S, Turel O, Li Y, Li J, Xue G, Chen A, He Q. Modulation of Brain Activity with Noninvasive Transcranial Direct Current Stimulation (tDCS): Clinical Applications and Safety Concerns. Front Psychol. 2017 May 10;8:685. doi: 10.3389/fpsyg.2017.00685. eCollection 2017. PMID 28539894
- [Background] Jahshan C, Rassovsky Y, Green MF. Enhancing Neuroplasticity to Augment Cognitive Remediation in Schizophrenia. Front Psychiatry. 2017 Sep 27;8:191. doi: 10.3389/fpsyt.2017.00191. eCollection 2017. PMID 29021765
- [Background] Matsumoto H, Ugawa Y. Adverse events of tDCS and tACS: A review. Clin Neurophysiol Pract. 2016 Dec 21;2:19-25. doi: 10.1016/j.cnp.2016.12.003. eCollection 2017. PMID 30214966
- [Background] Ekici B. Transcranial direct current stimulation-induced seizure: analysis of a case. Clin EEG Neurosci. 2015 Apr;46(2):169. doi: 10.1177/1550059414540647. No abstract available. PMID 25869110
- [Background] CANTAB® [Cognitive assessment software]. Cambridge Cognition (2019). All rights reserved. www.cantab.com
- [Background] Ruse SA, Harvey PD, Davis VG, Atkins AS, Fox KH, Keefe RS. Virtual Reality Functional Capacity Assessment In Schizophrenia: Preliminary Data Regarding Feasibility and Correlations with Cognitive and Functional Capacity Performance. Schizophr Res Cogn. 2014 Mar;1(1):e21-e26. doi: 10.1016/j.scog.2014.01.004. PMID 25083416
- [Background] Wilkinson, G. S., & Robertson, G. J. (2017). WRAT-5: Wide Range Achievement Test Professional Manual. Psychological Assessment Resources. https://books.google.ca/books?id=amQXtAEACAAJ
- [Background] Neil, S. T., Kilbride, M., Pitt, L., Nothard, S., Welford, M., Sellwood, W., & Morrison, A. P. (2009). The questionnaire about the process of recovery (QPR): A measurement tool developed in collaboration with service users. Psychosis, 1(2), 145-155. https://doi.org/10.1080/17522430902913450
- [Background] Faustman, W. O., & Overall, J. E. (1999). Brief Psychiatric Rating Scale. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment (p. 791-830). Lawrence Erlbaum Associates Publishers.
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Weissman AN, Beck AT. Development and validation of the dysfunctional Attitude Scale: A preliminary investigation. Paper presented at the Association for the Advancement of Behavior Therapy; Chicago. 1978.
- [Background] Fowler D, Freeman D, Smith B, Kuipers E, Bebbington P, Bashforth H, Coker S, Hodgekins J, Gracie A, Dunn G, Garety P. The Brief Core Schema Scales (BCSS): psychometric properties and associations with paranoia and grandiosity in non-clinical and psychosis samples. Psychol Med. 2006 Jun;36(6):749-59. doi: 10.1017/S0033291706007355. Epub 2006 Mar 27. PMID 16563204
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Cacioppo, J. T., & Petty, R. E. (1982). The need for cognition. Journal of Personality and Social Psychology, 42, 116-131.
- [Background] van der Gaag M, Schutz C, Ten Napel A, Landa Y, Delespaul P, Bak M, Tschacher W, de Hert M. Development of the Davos assessment of cognitive biases scale (DACOBS). Schizophr Res. 2013 Mar;144(1-3):63-71. doi: 10.1016/j.schres.2012.12.010. Epub 2013 Jan 15. PMID 23332365
- [Background] Llerena K, Park SG, McCarthy JM, Couture SM, Bennett ME, Blanchard JJ. The Motivation and Pleasure Scale-Self-Report (MAP-SR): reliability and validity of a self-report measure of negative symptoms. Compr Psychiatry. 2013 Jul;54(5):568-74. doi: 10.1016/j.comppsych.2012.12.001. Epub 2013 Jan 22. PMID 23351831
- [Background] Guleyupoglu B, Febles N, Minhas P, Hahn C, Bikson M. Reduced discomfort during high-definition transcutaneous stimulation using 6% benzocaine. Front Neuroeng. 2014 Jul 11;7:28. doi: 10.3389/fneng.2014.00028. eCollection 2014. PMID 25071548
- [Background] Kurzeck AK, Kirsch B, Weidinger E, Padberg F, Palm U. Transcranial Direct Current Stimulation (tDCS) for Depression during Pregnancy: Scientific Evidence and What Is Being Said in the Media-A Systematic Review. Brain Sci. 2018 Aug 14;8(8):155. doi: 10.3390/brainsci8080155. PMID 30110930